CLINICAL TRIAL: NCT06342557
Title: Integrated System for Patients Who Belong the Transition to Adult Services and Are Undergoing a Liver Transplant
Brief Title: Transitional ePRO Diary Liver
Acronym: MACROLIVER
Status: Recruiting | Type: Observational
Sponsor: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (Other)
Responsible Party: Sponsor
Other Study IDs: FROM
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Liver Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study is part of the MACROLIVER Project, whose main objective is to create a digital tool for patients and caregivers for the management of liver disease that allows the optimization of therapy and/or the treatment process, even remotely. Such a tool not only reduces the movement of patients who are by definition fragile, but also enables the optimization of access and care by a multidisciplinary team. This tool is intended to support doctors and patients, but in no way replaces normal clinical practice. This study aims to explore the specificities of patients experiencing the transition from the pediatric ward to the adult ward in order to identify risk and protective factors that influence psychological well-being at both an individual and relational level. In order to gather all the information about the patients attending the transitional clinic and to obtain a more complete and truthful clinical-psychological picture, the study also includes the collection of retrospective data of the transplanted patients.

ELIGIBILITY:
Inclusion Criteria:

* patients between the ages of 14 and 20 who have been transplanted at the ASST-PG23 transplant center or are awaiting a liver transplant and belong to the transition to adult services
* signed informed consent
* proven use of the APPs (to be assessed based on the last 2 weeks)

Exclusion Criteria:

-

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients between the ages of 14 and 20 who have been transplanted at the ASST-PG23 transplant center or are awaiting a liver transplant and belong to the transition to adult services.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2034-02-21 (Estimated); Study Completion 2034-02-21 (Estimated)

PRIMARY OUTCOMES:
four-item Morisky Medication Adherence Scale (MGLS) | 3 months
  MGLS is used to assess non-adherence to therapy. The MGLS includes four questions with yes/no response options, resulting in a score from 0 to 4. Based on this score, there are 3 levels of adherence: high, medium and low adherence with 0, 1-2 and 3-4 points respectively. Scores below 2 indicate a lack of adherence to therapy, while scores greater than or equal to 3 indicate adherence to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Fagiuoli, MD, Principal Investigator — ASST-PG23
Locations (1):
- ASST-Papa Giovanni XXIII, Bergamo, MILANO, Italy

IPD SHARING:
Plan to Share IPD: No